CLINICAL TRIAL: NCT02769897
Title: Obesity in Schoolchildren of Basic Education: a Study of Interdisciplinary Intervention - Phase III
Brief Title: Obesity in Schoolchildren of Basic Education - Phase III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santa Cruz do Sul (Other)
Responsible Party: Principal Investigator, Miria Suzana Burgos, Dr, University of Santa Cruz do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 54985316.0.0000.5343
Record Dates: First submitted 2016-05-06; First posted 2016-05-12 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Obesity; Adolescent Behavior
MeSH Terms: conditions — Obesity; Adolescent Behavior | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): The exercise program, nutritional counseling and oral health will last for five to six months and will be held in the gym and rooms of the University of Santa Cruz do Sul (UNISC). The sessions will last two hours (one hour of physical exercise and the second time divided into nutritional counseling, postural, psychological and oral) with a frequency of three times a week.
  Interventions: Behavioral: Physical exercise
- Control group (No Intervention): The control group did not receive the intervention.

INTERVENTIONS:
Behavioral: Physical exercise — The sessions will last two hours (one hour of physical exercise and the second time divided into nutritional counseling, postural, psychological and oral) with a frequency of three times a week.
  Other Names: Nutritional counseling
  Arms: Intervention group

SUMMARY:
The study aims to evaluate the possible effects of an exercise program, nutritional and psychological, postural orientation and guidance of oral health on body composition, physical activity levels and lifestyle, physical fitness and health and motor performance, the factors risk of cardiovascular disease, eating habits, the cognition levels, the psychological profile, the body posture of children and adolescents with overweight and obesity, considering the presence of risk genotype associated with the development of obesity. In addition, identify the effects of orientation for oral health on the quality of life and healthy oral habits.

DETAILED DESCRIPTION:
The study aims to evaluate the possible effects of an exercise program, nutritional and psychological, postural orientation and guidance of oral health on body composition, physical activity levels and lifestyle, health-related physical fitness and motor performance in factors risk of cardiovascular disease, eating habits, cognition levels, psychological profile and body posture of adolescents with overweight and obesity. In addition, identify the effects of orientation for oral health on the quality of life and healthy oral habits. A quasi-experimental research will consist of a sample of approximately fifty adolescents with overweight and obesity, ages 10 to 17, of both sexes, selected voluntarily in two schools in Santa Cruz do Sul. The sessions will last two hours (one hour of physical exercise and the second time divided into nutritional counseling, postural, psychological and oral orientation) with a frequency of three times a week. The exercise session will consist of 10 minutes of warm-ups, 40 minutes of aerobic exercise, recreational and sports activities (moderate to severe) and 10 minutes back to calm, and the intensity of the activities will be monitored through a frequency (target heart rate: 60 to 70% of maximum heart rate of each subject). Nutritional, psychological, postural and oral guidance will be given by a nutritionist, psychologist, physiotherapist/physical education professional and odontologist respectively, which present lectures and educational games. The following parameters will be evaluated: anthropometric (BMI, waist circumference and skinfold thickness); hematologic and biochemical analysis (HDL cholesterol, LDL cholesterol, total cholesterol, triglycerides, glucose, insulin, adiponectin, leptin, resistin, C reative protein, ALT, AST, glycated hemoglobin, IL-6, IL-10, TNF-α, cortisol, irisina, F2 isoprostane and uric acid); polymorphism related to obesity (FTO rs9939609); related-health physical fitness (flexibility; sit and reach test; abdominal strength and cardiorespiratory fitness); postural deviations evaluated by the photogrammetry method - SAPO program. The nutritional habits and lifestyle will be assessed by self-report a validated and adapted questionnaire for Brazilian children and adolescents as well as a recall and diet calculation for nutrients through Virtual Nutri 1.0. Oral health will be evaluated according to the criteria of the SB Brazil Project 2010. The psychological and cognitive assessment will be done through instruments that determine self-esteem, body awareness, stress and possible mental health problems of adolescent. The results will be presented by means of statistical tests performed using SPSS 23.0. The comparison of the average values of variables between pre- and post-intervention will be carried out through the Anova test for repeated measures (generalized linear models), with subsequent calculation of the effect size; the two-way ANOVA is used to analyze the differences among the changes in the control group and the experimental group. Expected results: It is expected that after the completion of this research project, there are increases in the levels of cardiorespiratory fitness, flexibility and abdominal strength, changes in postural deviations and dietary habits, increased cognitive function and psychological aspects and improved hygiene and perception of oral health of adolescents with overweight and obesity and consequent reduction in rates of overweight and obesity and the risk factors of cardiovascular disease. The aim is to collaborate with public health policies in the prevention and treatment of overweight and obesity and consequences in schools.

ELIGIBILITY:
Inclusion Criteria:

* The official signing the informed consent and informed;
* The student with 12 years or older must sign the consent term;
* Age range: 10 to 17years;
* Gender: male and female;
* No contraindications for blood collection;
* No distinction in relation to social class, ethnicity or color;
* To have a BMI greater than 85th percentile;
* Do not be participating in any other exercise program and dietary intervention;
* Participate in the clarification meetings on the project, when the head of the student is committed to the project, the following: a) assume responsibility for bringing to the UNISC (building 42) and refer to their home, the participant student of this study, both in the days of assessment (testing and completion of the data collection instruments), as in the days of intervention: 2nd, 4th and 6th fairs, from 14h to 16h, including 15 minutes in advance to the host, call and guidance students;
* Participate in intervention sessions during the period of 2 hours daily, the established days, following the guidelines given by the coordination of the project and the professionals of Physical Education, Nutrition, Psychology, Pharmacy, Physiotherapy, Medicine, Nursing and / or another area of health / education that can contribute to achieving the objectives of the intervention project;
* Participate in the assessments and reassessments as protocols established by the project.

Exclusion Criteria:

* Students who submit a frequency less than 70% stake in the intervention;
* Students who present contraindication to the practice of physical activity during the program implementation period;
* Students who choose not to continue with the treatment of intervention proposed by the program;
* Be in possession of any kind of illness, abnormality or health problem such as: Hypertension untreated, Kidney diseases, Cardiac disorders, chronic renal failure, genetic diseases that have congenital malformations and mental retardation as Turner syndrome, Klinefelter syndrome and Down syndrome or cognitive impairment. And do not be carrying transmitted diseases vertically (from mother to child) with anatomical deformations caused by the interference of the pathogenic agent in the development process, as Congenital Toxoplasmosis (hydrocephalus, cerebral calcification, mental retardation, acute myocarditis, retinochoroiditis, strabismus, microphthalmia ), Rubella Syndrome, congenital (deafness, congenital cataracts, heart defects, microcephaly and mental retardation) congenital Syphilis (bone deformities, keratitis, deafness and mental retardation), cytomegalovirus infection congenital (microcephaly, intracranial calcifications and sensorineural deafness), because these subjects they need special care medical and/or service people trained for the specific purposes.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Body mass index (kg/m²) | 6 months
  Body mass index is measured by the weight and height values, applying the formula: weight/(height)²

IPD SHARING:
Plan to Share IPD: Undecided
The results will be submitted to scientific journals.